CLINICAL TRIAL: NCT02207335
Title: A Multicenter Randomized Phase Ⅲ Clinical Trial of Gemcitabine in Combination With Capecitabine Versus Gemcitabine Plus Carboplatin as First-line Treatment in Triple-negative Recurrent or Metastatic Breast Cancer
Brief Title: Trial of Gemcitabine_Capecitabine Versus Gemcitabine_Carboplatin in Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIH-TZS-20140421-01
Record Dates: First submitted 2014-04-22; First posted 2014-08-04 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2013-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine，Capecitabine (Experimental): Gemcitabine: 1250 mg/m2, ivgtt, 30mins, D1,8 Capecitabine: 1250 mg/m2, PO, Q12h, D1-14
  Interventions: Drug: Gemcitabine，Capecitabine
- Gemcitabine, Carboplatin (Active Comparator): Gemcitabine: 1250 mg/m2, ivgtt,30mins, D1,8 Carboplatin: AUC 2, ivgtt, 60mins, D1,8
  Interventions: Drug: Gemcitabine, Carboplatin

INTERVENTIONS:
Drug: Gemcitabine，Capecitabine — Gemcitabine: 1250 mg/m2, ivgtt, 30mins, D1,8 Capecitabine: 1250 mg/m2, PO, Q12h, D1-14
  Arms: Gemcitabine，Capecitabine
Drug: Gemcitabine, Carboplatin — Gemcitabine: 1250 mg/m2, ivgtt,30mins, D1,8 Carboplatin: AUC 2, ivgtt, 60mins, D1,8
  Arms: Gemcitabine, Carboplatin

SUMMARY:
Gemcitabine plus carboplatin in recurrent or metastatic breast cancer is a recommended scheme in National Comprehensive Cancer Network (NCCN) guideline. gemcitabine in combination with capecitabine is also effective in Metastatic Breast Cancer (MBC) in some clinical study with small sample.

DETAILED DESCRIPTION:
A multicenter randomized phase Ⅲ clinical trial of gemcitabine in combination with capecitabine versus gemcitabine plus carboplatin as first-line treatment in triple-negative recurrent or metastatic breast cancer.The primary endpoints of the study is progression free survival (PFS). The secondary endpoints are overall response rate (ORR), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-70 years old
* ECOG 0-1
* Expected lifetime more than 12 weeks

Exclusion Criteria:

* Pregnancy
* Brain Metastasis,
* Severe Infection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
RECIST 1.1 | -7 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhongsheng Tong, Master, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Liu X, Zhao W, Jia Y, Shi Y, Wang X, Li S, Zhang P, Wang C, Hao C, Tong Z. A non-inferiority, phase III trial of gemcitabine plus capecitabine versus gemcitabine plus carboplatin as first-line therapy and tumor-infiltrating lymphocytes as a prognostic biomarker in patients with advanced triple-negative breast cancer. Ther Adv Med Oncol. 2024 Dec 3;16:17588359241240304. doi: 10.1177/17588359241240304. eCollection 2024. PMID 39634173
- [Derived] Egger SJ, Chan MMK, Luo Q, Wilcken N. Platinum-containing regimens for triple-negative metastatic breast cancer. Cochrane Database Syst Rev. 2020 Oct 21;10(10):CD013750. doi: 10.1002/14651858.CD013750. PMID 33084020